CLINICAL TRIAL: NCT05877352
Title: Intraoperative Electron Radiotherapy in Rectal Cancer - A Feasibility Trial
Acronym: ELECTRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: IntraOp Medical Corporation (Unknown); PLANETS Cancer Charity (Unknown); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RHMCAN1600; ISRCTN48105173 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2023-03-29; First posted 2023-05-26 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Rectal Cancer; Locally Recurrent Rectal Cancer

STUDY DESIGN:
Intervention Model Description: A single centre double-blinded three-arm randomised controlled trial of extended margin surgery + IOERT at standard dose (10 Gy) versus extended margin surgery + IOERT at higher dose (15 Gy) versus extended margin surgery alone (no IOERT) in a 1:1:1 ratio in patients with LARC or LRRC.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blinded trial, which means both the participant and clinicians will not know the treatment allocation. The surgeon, oncologist and patient will remain blinded throughout the study, while the radiotherapy delivery team will know the outcome of the randomisation.
  Patient allocation will be provided to the unblinded radiotherapy staff via an Interactive Web Response System (IWRS). The randomisation code will be retained by the system. Deaths and serious adverse events (SAE) will be reviewed in a blinded manner.
  Unblinding will be required in the event that any participants further treatment may benefit from further radiotherapy, and if potential IOERT treatment and its dose may impact this.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No IOERT (Active Comparator): Extended margin surgery
  Interventions: Procedure: Extended Margin Surgery
- Low Dose IOERT (Experimental): Extended margin surgery and IOERT at standard dose (10 Gy)
  Interventions: Radiation: Intraoperative Electron Radiotherapy (IOERT); Procedure: Extended Margin Surgery
- High Dose IOERT (Experimental): Extended margin surgery and IOERT at higher dose (15 Gy)
  Interventions: Radiation: Intraoperative Electron Radiotherapy (IOERT); Procedure: Extended Margin Surgery

INTERVENTIONS:
Radiation: Intraoperative Electron Radiotherapy (IOERT) — IOERT can be defined as the direct application of high-energy electron beam irradiation to a tumour bed during an operative procedure. This approach permits precise delivery of a single large fraction of radiation directly and specifically to high recurrence risk anatomical target areas, which the treating clinicians (surgeon and attending clinical oncologist) predict will be a close or involved margin, while simultaneously displacing and shielding dose-limiting radiosensitive structures such as the small bowel or ureter or any anastomoses, if not involved by tumour.
  Arms: High Dose IOERT; Low Dose IOERT
Procedure: Extended Margin Surgery — Surgery intended to remove both a tumour and any metastases

SUMMARY:
Single centre double-blinded three-arm randomised controlled trial of extended margin surgery + IOERT at standard dose (10 Gy) versus extended margin surgery + IOERT at higher dose (15 Gy) versus extended margin surgery alone in a 1:1:1 ratio in patients with Locally Advanced Rectal Cancer (LARC) or Locally Recurrent Rectal Cancer (LRRC).

DETAILED DESCRIPTION:
Rectal cancer is a cancer that occurs in the pelvis from the rectum. Locally advanced rectal cancer outgrows the rectum and attaches to other body parts in the pelvis and locally recurrent rectal cancer is a rectal cancer that comes back after surgery, and usually attaches to many different pelvic structures. They are both difficult to manage. The standard of care treatment involves chemotherapy and radiotherapy, followed by what is known as an extended margin operation to remove all cancer affected organs and not leave any cancer cells behind. If cancer cells reach the edge of the removed tissue, there is a high chance of leaving cancer cells behind. This is a key predictor of negative outcome in patients. Intraoperative electron beam radiotherapy (IOERT) was developed to help improve patient outcomes. Once the cancer has been removed, the surgeon and a cancer radiotherapy specialist examine the patient's scans, the cancer specimen and the area the cancer was in, and if there is concern about small numbers of cancer cells being left behind they treat the area with radiotherapy to destroy these cells. Patients that are due to receive treatment for these subsets of rectal cancer will be approached to take part. If eligible on the day of surgery the patient will be randomised to one of three arms: Arm A - standard of care (No IOERT), Arm B - extended margin surgery plus IOERT (10 Gy), or Arm C - extended margin surgery plus higher dose IOERT (15 Gy). The surgeon, cancer specialist team and patient will be blinded to study treatment. Patients will be followed up at 30 days, 3 months and for a minimum of 12 months post surgery as part of the trial and they will be followed up for 5 years as part of standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16
* Non-metastatic/oligo-metastatic (up to 3 lesions from 2 sites predicted to be radically treatable) - locally advanced or locally recurrent disease involving the posterior or lateral components of the pelvis and predicted to be resectable but with close margins from imaging as determined by a specialist MDT (sMDT)
* Colorectal sMDT review with experience in pelvic exenteration, which has proposed IntrOperative Electron Radiotherapy (IOERT) as an option for treatment
* Patient suitable for IOERT as component of treatment in the view of the responsible Clinical Oncologist
* Performance status ≤1 as defined by the Eastern Cooperative Oncology Group (ECOG)
* Deemed medically fit for surgery
* Written informed consent

Exclusion Criteria:

* Unresectable disease/likelihood of R2 resection
* sMDT determined excess prior radiotherapy within IOERT target zone
* Women who are pregnant or breastfeeding
* Participation within an interventional clinical trial within 3 months of the point of registration within ELECTRA

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Patients meeting eligibility criteria | 2 years
  Number and percentage of patients meeting eligibility criteria and number of patients referred to a sMDT over the trial period
Patients accepting randomisation | 2 years
  Number and percentage of patients accepting randomisation
Successful delivery of IOERT | 2 years
  Number and percentage of patients for which IOERT was successfully delivered as planned as part of the trial
Blind maintained for patients and clinicians | 2 years
  Number and percentage of patients and clinicians for which blinding was maintained for IOERT delivery
Questionnaire analysis | 2 years
  Percentage of patients whose questionnaires can be analysed
Availability of potential primary outcome data | 2 years
  Percentage of patients for whom we can collect information on potential primary outcomes

SECONDARY OUTCOMES:
Morbidity | Up to 30 days post randomisation
  Clavien Dindo classification
Mortality | 30 days post randomisation
  Mortality
IOERT Field Recurrence | 12 months post randomisation
  IOERT Field Recurrence is defined as the area directly within the IOERT field as marked by ligaclips or identified by the surgical oncologist for future radiological surveillance.
Overall local recurrence | 12 months post randomisation
  Overall local recurrence (OLR) is defined as including both IOERT-field and non-IOERT field loco-regional recurrences.
Overall survival | 12 months post randomisation
  Overall survival
Treatment related toxicity | 12 months post randomisation
  Treatment related toxicity graded by CTCAE v5
Time to local or systemic recurrence | Time from randomisation to local or systemic recurrence or 3 years post the start of recruitment, whichever comes first
  Time to local or systemic recurrence
R1 Rate | At randomisation
  R1 Rate
EQ-5D-5L | At 3 and 12 months post randomisation
  Quality of life scored from EQ-5D-5L
LRRC QoL | At 3 and 12 months post randomisation
  Quality of life scored from LRRC QoL
QLQ-C30 | At 3 and 12 months post randomisation
  Quality of life scored from QLQ-C30
SF-36 | At 3 and 12 months post randomisation
  Quality of life scored from SF-36
Resource use and cost | At 3 and 12 months post randomisation
  Cost will be estimated for the NHS. An NHS and social care perspective will be used, including intervention costs, outpatient visits and investigations, A&E attendances, hospital admissions, number and dose of each radiotherapy treatment. Itemised resource usage date will be priced using appropriate national sources: Personal Social Services Research Unit (PSSRU), NHS Reference costs and BNF (British National Formulary) for the UK.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Mirnezami, Prof, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No